CLINICAL TRIAL: NCT02002221
Title: A 12-week, Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Equa (Vildagliptin) 50 mg Bid as an add-on Therapy to Insulin, With or Without Metformin, in Patients With Type 2 Diabetes Mellitus
Brief Title: Study of Efficacy and Safety of Vildagliptin as add-on Insulin Therapy in T2DM Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A1405
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes Mellitus (DM) ,; diabetes,; noninsulin-dependent diabetes mellitus (NIDDM),; adult-onset diabetes,; high blood sugar,; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; Insulin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Vildagliptin (LAF237) (Experimental): Patients received vildagliptin (LAF237) 50 mg tablets twice daily for 12 weeks. Patients continued on a stable dose of long-acting or intermediate-acting or pre-mixed insulin, and metformin if applicable, throughout the study
  Interventions: Drug: Vildagliptin (LAF237); Drug: Insulin; Drug: Metformin
- Placebo (Placebo Comparator): In this arm, patients received vildagliptin 50 mg matching placebo tablets twice daily for 12 weeks. Patients continued on a stable dose of long-acting or intermediate-acting or pre-mixed insulin, and metformin if applicable, throughout the study
  Interventions: Drug: Placebo; Drug: Insulin; Drug: Metformin

INTERVENTIONS:
Drug: Vildagliptin (LAF237) — Corresponds to vildagliptin (LAF237) 50 mg tablets twice daily
  Other Names: Vildagliptin
  Arms: Vildagliptin (LAF237)
Drug: Placebo — Matching placebo of vildagliptin 50 mg twice daily
  Arms: Placebo
Drug: Insulin — Patients continued their prescribed insulin dose. The dose of insulin remained within a 10% increase of the baseline dose throughout the trial (with no change in frequency or insulin type) unless dose adjustments were required for safety reasons.
  The insulin dose was allowed to be decreased for safety reasons at anytime without specific dose limits at the Investigator's discretion.
Drug: Metformin — Patients continued their prescribed metformin dose, if applicable.

SUMMARY:
The purpose of this study was to assess the efficacy and safety of vildagliptin 50 mg bid add-on therapy to improve overall glycemic control in patients with T2DM inadequately controlled by insulin, with or without concomitant metformin treatment. It was agreed with PMDA to conduct a postmarketing clinical trial to further collect the efficacy and safety data of vildagliptin especially in Japanese patients when it iwas used on top of insulin.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of T2DM by standard criteria.
* HbA1c ≥ 7.0 to ≤ 10% at Visit 1.
* Age: ≥ 20 to < 75 years old at Visit 1.
* BMI ≥ 20 to ≤ 35 kg/m2 at Visit 1.

Exclusion Criteria:

* FPG ≥ 270 mg/dL (≥15 mmol/L) at Visit 1.
* Type 1 diabetes, monogenic diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes.
* Significant heart diseases
* Hepatic disorder

Other protocol defined inclusion/exclusion criteria may apply

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Japan (25):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukutsu, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Ibusuki, Kagoshima-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Yatsushiro, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Ageo, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Adachi-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Suginami-ku, Tokyo

REFERENCES:
- [Derived] Hirose T, Suzuki M, Tsumiyama I. Efficacy and Safety of Vildagliptin as an Add-on to Insulin with or without Metformin in Japanese Patients with Type 2 Diabetes Mellitus: A 12-week, Double-Blind, Randomized Study. Diabetes Ther. 2015 Dec;6(4):559-571. doi: 10.1007/s13300-015-0147-6. Epub 2015 Nov 30. PMID 26620049

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vildagliptin (LAF237) | Placebo
Started | 78 | 78
Completed | 76 | 75
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Patient withdrew consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vildagliptin (LAF237) | Placebo | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.5 (9.57) | 60.1 (9.11) | 59.3 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 55 | 56 | 111

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 12 Weeks Between Treatment Groups
Description: HbA1c was performed on a blood sample obtained and measured by high performance liquid chromatography performed at a central laboratory.
Time Frame: Baseline, week 12
Population: The full analysis set consisted of all randomized patients who received at least one dose of study medication and had at least one post-baseline assessment of efficacy parameter measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Vildagliptin (LAF237) | Placebo
Number analyzed (Participants) | 78 | 78
percentage of glycosylated haemoglobin | -1.01 (0.06) | -0.11 (0.06)
Statistical Analysis 1: Comparison: Vildagliptin (LAF237) vs Placebo; H0: δ vildagliptin 50 mg bid = δ placebo versus H1: δ Vildagliptin 50 mg bid < δ placebo,; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.91, 95% CI 2-sided [-1.08 to -0.73], Standard Error of Mean 0.09

2. Secondary Outcome: Percentage of Patients Meeting Responder Rates in HbA1c
Description: Responder rate was analyzed in categories: Criterion 1- Endpoint HbA1c ≤ 6.5%, Criterion 2- Endpoint HbA1c < 7% , Criterion 3- Endpoint HbA1c < 7% in patients with baseline HbA1c ≤ 8%, Criterion 4- HbA1c reduction from baseline at endpoint ≥ 1%, Criterion 5- HbA1c reduction from baseline at endpoint ≥ 0.5%. The number of patients analyzed for Criterion 1 and 2 include only patients with baseline HbA1c ≥ 7% (> 6.5%) and endpoint HbA1c measurement. The number of patients analyzed for Criterion 3 includes only patients with 7% ≤ baseline HbA1c ≤ 8% and endpoint HbA1c measurement. The number of patients analyzed for Criterion 4 and 5 include patients with both baseline and endpoint HbA1c measurements.
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Vildagliptin (LAF237) | Placebo
Number analyzed (Participants) | 78 | 78
percentage of patients
  At least one criterion met (n = 78, 78) | 67 | 21
  Criterion 1 (n= 77, 78) | 23 | 2
  Criterion 2 (n= 76, 77) | 38 | 3
  Criterion 3 (n= 42, 37) | 33 | 3
  Criterion 4 (n=78, 78) | 38 | 5
  Criterion 5 (n= 78, 78) | 62 | 20

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at 12 Weeks
Description: FPG was performed on a blood sample obtained and analyzed at a central laboratory.
Time Frame: Baseline, week 12
Population: The full analysis set consisted of all randomized patients who received at least one dose of study medication and had at least one post-baseline assessment of efficacy parameter measurement. Number of patients with observations at both baseline and endpoint are analyzed in this endpoint.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Vildagliptin (LAF237) | Placebo
Number analyzed (Participants) | 78 | 78
mg/dL | -21.87 (4.05) | -0.30 (4.04)

4. Secondary Outcome: Number of Participants With Incidence of Hypoglycemia and Severe Hypoglycemia
Description: Hypoglycemic events are defined as a) symptoms suggestive of hypoglycemia, where the patient is able to initiate self-treatment and plasma glucose measurement is < 56 mg/dL (grade 1), b) symptoms suggestive of hypoglycemia, where the patient is unable to initiate self-treatment and plasma glucose measurement is < 56 mg/dL (grade 2), c) symptoms suggestive of hypoglycemia, where the patient is unable to initiate self-treatment and no plasma glucose measurement is available (suspected grade 2)
Time Frame: 12 weeks
Population: The safety set consisted of all patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Vildagliptin (LAF237) | Placebo
Number analyzed (Participants) | 78 | 78
Participants
  at least one hypoglycemic event | 5 | 1
  grade 2 hypoglycemic events | 0 | 0
  suspected grade 2 hypoglycemic events | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death
Description: The occurrence of adverse events was sought by non-directive questioning of the patient at each visit. Adverse events are defined as appearance or worsening of any undesirable symptom, vital sign, or medical conditions. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: 12 weeks
Population: The safety set consisted of all patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Vildagliptin (LAF237) | Placebo
Number analyzed (Participants) | 78 | 78
Participants
  Any adverse events | 36 | 34
  Serious adverse events | 2 | 1
  Death | 0 | 0

ADVERSE EVENTS:
Description: The safety set consisted of all patients who received at least one dose of study medication. Patients were analyzed according to the treatment received.
Arm/Group | Vildagliptin (LAF237) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/78 | 1/78
Other Adverse Events (participants affected / at risk) | 22/78 | 21/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin (LAF237) (N=78) | Placebo (N=78)
Angina pectoris (Cardiac disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin (LAF237) (N=78) | Placebo (N=78)
Asthenia (General disorders) | 6 | 6
Hunger (General disorders) | 7 | 3
Nasopharyngitis (Infections and infestations) | 10 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 1
Tremor (Nervous system disorders) | 7 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.